CLINICAL TRIAL: NCT02796053
Title: Study to Assess Pharmacodynamics, Clinical Effects, Safety and Pharmacokinetics of TAB08 in Patients With Psoriasis Vulgaris, Not Adequately Controlled With Current Concomitant Therapy
Brief Title: TAB08 in Patients With Psoriasis Vulgaris, Not Adequately Controlled With Current Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Theramab LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAB08-PSO-01
Record Dates: First submitted 2016-05-24; First posted 2016-06-10 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — TGN-1412

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo to TAB08
  Interventions: Other: Placebo
- TAB08 Dose 1 (Experimental): Drug: TAB08 biologic
  Interventions: Drug: TAB08

INTERVENTIONS:
Drug: TAB08 — The TAB08 will be administered intravenously, by infusion.
  Arms: TAB08 Dose 1
Other: Placebo — The Placebo to TAB08 will be administered intravenously, by infusion.
  Arms: Placebo

SUMMARY:
Study to assess Pharmacodynamics, Safety, Pharmacokinetics and clinical effects of TAB08 during 12 weeks of treatment in patients with Psoriasis Vulgaris, not adequately controlled with current therapy.

DETAILED DESCRIPTION:
1. To assess dynamics of the T-lymphocytes subpopulations in patients peripheral blood during 12 weeks of TAB08 treatment.
2. To assess dynamics of selected cytokines levels in patients peripheral blood during 12 weeks of TAB08 treatment.
3. To assess TAB08 concentrations in patients blood during 12 weeks of TAB08 treatment.
4. To assess frequency, seriousness and severity of adverse events during 12 weeks of TAB08 treatment.
5. To assess changes in PASI, IGA and DLQI during 12 weeks of TAB08 treatment and subsequent 4 weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Vulgar Psoriasis
* Area of Psoriasis skin damage ≥ 10%
* PASI Score ≥ 12
* Score on IGA scale ≥ 3

Exclusion Criteria:

* Other forms of psoriasis in addition to vulgar
* Prohibited treatment
* Pregnant or nursing women
* Concomitant systemic therapy dosage modification (if any) within 4 weeks before randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change of T-lymphocytes subsets in absolute count (number of cells per mL) in peripheral blood at Weeks 2, 3, 4, 8 and 12 comparing to Baseline. | 12 weeks
Change of T-lymphocytes subsets (in percent) in peripheral blood at Weeks 2, 3, 4, 8 and 12 comparing to Baseline. | 12 weeks
Change of cytokines concentrations (in micrograms/mL) in peripheral blood at Weeks 2, 3, 4, 8 and 12 comparing to Baseline. | 12 weeks
Change of cytokines concentrations (in percent) in peripheral blood at Weeks 2, 3, 4, 8 and 12 comparing to Baseline. | 12 weeks

SECONDARY OUTCOMES:
TAB08 concentrations in peripheral blood | 12 weeks
Adverse events frequency, seriousness and severity | 16 weeks
Psoriasis Area Severity Index (PASI) | 16 weeks
Investigator Global Assessment (IGA) | 16 weeks
Patient-reported health outcome assessed by Short Form - Dermatology Quality of Life Index (DLQI) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniil Nemenov, M.D., Study Director — Theramab LLC
Locations (1):
- Clinical Emergency Hospital of Yaroslavl, Yaroslavl, Russia

IPD SHARING:
Plan to Share IPD: Undecided